CLINICAL TRIAL: NCT02635178
Title: Randomized Control Trial Examining a Brief Anxiety Sensitivity Cognitive Concerns Intervention for Obsessive Compulsive Symptoms
Brief Title: Brief Anxiety Sensitivity Treatment for Obsessive Compulsive Symptoms
Acronym: COAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Raines02
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Obsessive-Compulsive Disorder and Symptoms
Keywords: Obsessive-compulsive disorder; OCD; Anxiety sensitivity; Cognitive Concerns
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Cognitive Anxiety Sensitivity Treatment (CAST) is a computerized treatment designed to model the educational and behavioral techniques used in anxiety treatments. The psychoeducational component focuses on the nature of stress and its effects on the mind and body. CAST was designed to dispel myths concerning the immediate dangers of stress on cognitive processes. Individuals are taught that psychological arousal from stress is not dangerous and that they may have developed a conditioned fear to these sensations, as indicated by their elevated levels of AS cognitive concerns. In addition to psychoeducation, interoceptive exposure exercises will be introduced to correct the conditioned fear response. The program will demonstrate exercises that elicit sensations consistent with AS cognitive concerns.
  Interventions: Behavioral: Cognitive Anxiety Sensitivity Treatment
- Control (Placebo Comparator): The Physical Health Education Training (PHET) control condition was designed to control for the effects of general education provided in the CAST condition. Participants will be presented with information regarding the importance and benefits of maintaining a healthy lifestyle. The program will discuss diet, alcohol and water consumption, exercise, sexual health, and sleep. PHET will instruct the participant how to monitor their daily health habits in order to achieve a healthy lifestyle. PHET will take approximately 45 minutes to complete. Based on the findings of Schmidt and colleagues (in press), this intervention does not appear to exert a strong effect on AS.
  Interventions: Behavioral: Physical Health Education Training

INTERVENTIONS:
Behavioral: Cognitive Anxiety Sensitivity Treatment — Cognitive Anxiety Sensitivity Treatment (CAST) is a computerized treatment designed to model the educational and behavioral techniques used in anxiety treatments. The psychoeducational component focuses on the nature of stress and its effects on the mind and body. CAST was designed to dispel myths concerning the immediate dangers of stress on cognitive processes. Individuals are taught that psychological arousal from stress is not dangerous and that they may have developed a conditioned fear to these sensations, as indicated by their elevated levels of AS cognitive concerns. In addition to psychoeducation, interoceptive exposure exercises will be introduced to correct the conditioned fear response. The program will demonstrate exercises that elicit sensations consistent with AS cognitive concerns.
  Arms: Active
Behavioral: Physical Health Education Training — The Physical Health Education Training (PHET) control condition was designed to control for the effects of general education provided in the CAST condition. Participants will be presented with information regarding the importance and benefits of maintaining a healthy lifestyle. The program will discuss diet, alcohol and water consumption, exercise, sexual health, and sleep. PHET will instruct the participant how to monitor their daily health habits in order to achieve a healthy lifestyle. PHET will take approximately 45 minutes to complete. Based on the findings of Schmidt and colleagues (in press), this intervention does not appear to exert a strong effect on AS.
  Arms: Control

SUMMARY:
Obsessive-compulsive disorder (OCD), characterized by recurrent obsessions and/or compulsions, is a disabling psychiatric condition affecting approximately 2-3% of the population. Whereas several first-line treatments have been established (e.g., pharmacological and psychological), a substantial proportion of patients (40-60%) fail to experience symptom remission, underscoring the need for research in this area. One approach to increasing treatment efficacy is to target underlying risk factors or dysfunctions that may in turn improve outcomes. One such risk factor is anxiety sensitivity (AS) cognitive concerns. AS cognitive concerns reflects fears of mental incapacitation (e.g., "It scares me when I am unable to keep my mind on a task"). There is recent evidence that AS cognitive concerns is uniquely associated with various obsessive-compulsive (OC) symptom domains. However, questions remain as to whether reductions in AS cognitive concerns will lead to subsequent reductions in OC symptoms. The purpose of the proposed study is to investigate the efficacy of a brief AS cognitive concerns intervention on reductions in OC symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Elevated levels of obsessive-compulsive symptoms as indicated by scoring one standard deviation above the non-clinical mean on any Dimensional Obsessive-Compulsive Scale dimension
* Elevated anxiety sensitivity cognitive concerns as indicated by scoring one standard deviation above the non-clinical mean

Exclusion Criteria:

* Evidence of a significant medical illness that would prevent the completion of interoceptive exposure (IE) exercises
* Non-English speakers
* Individuals currently receiving cognitive-behavioral therapy for anxiety and/or mood disorders or who are not stable on psychotropic medications (i.e., new medication or changes in dosage within the last three months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index-3 (ASI-3) | Month 1 Follow-Up
  The ASI-3 is an 18-item self-report measure of AS. This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the original ASI provides. The measure has shown good psychometric properties (Taylor et al., 2007).

SECONDARY OUTCOMES:
Dimensional Obsessive Compulsive Scale (DOCS) | Month 1 Follow-Up
  The DOCS is a 20-item measure that assesses the four dimensions of OC symptoms most reliably replicated in previous structural research. This measure includes four subscales: contamination, responsibility, unacceptable thoughts, and symmetry. The DOCS demonstrates excellent psychometric properties and has been validated in both clinical and non-clinical samples (Abramowitz et al., 2010).
Sheehan Disability Scale (SDS) | Month 1 Follow-Up
  The SDS is a 3-item self-report measure designed to assess functional impairment in work/school, social, and family life. The measure has shown good psychometric properties (Sheehan et al., 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M Raines, M.S., Principal Investigator — Florida State University

IPD SHARING:
Plan to Share IPD: No
Members of the scientific community can request a copy of the data by contacting the PI, Amanda Raines. They should state their reason for request and plans for analyzing. A limit dataset would be created, encrypted, and sent.